CLINICAL TRIAL: NCT02485132
Title: Evaluating the True Magnitude of HYPOglycemic Events After THE Initiation of Sulfonylurea, by Continuous Glucose monItoring System: A Multicenter Study. The HYPOTHESIS Trial
Brief Title: Evaluating the True Magnitude of HYPOglycemic Events After THE Initiation of Sulfonylurea
Status: Terminated | Type: Observational
Why Stopped: Patients corresponding to the inclusion/exclusion criteria not found.
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Other Study IDs: HYPOTHESIS
Record Dates: First submitted 2015-06-21; First posted 2015-06-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Sulfonylurea; Hypoglycemia; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- T2DM at SU initiation: T2DM newly prescribed a SU
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Investigators propose to perform a one-week baseline testing (pre-initiation of the SU), at initiation (first week after the first dose of the SU) and after a 3 months follow-up of treatment with a SU, including CGMS reading, medical history measures, quality of life and diabetes treatment satisfaction.

SUMMARY:
Sulfonylurea are known to be associated with a risk of hypoglycaemia. However, little is known about the real frequency of asymptomatic or unreported hypoglycemia and their impact on glycemic control and quality of life among patients using sulfonylureas (SUs). The frequency of hypoglycemia is probably underestimated since self-monitoring of blood glucose (SMBG) fail to identify asymptomatic episodes, especially among patients with higher risk of hypoglycemia unawareness (longer diabetes duration, elderly, recurrent hypoglycemia, etc.). No previous studies have reported total hypoglycemia as measured by continuous glucose monitoring system (CGMS) in a large group of Canadians, therefore underestimating the true incidence of these events. As with age hypoglycemia perception is reduced and consequences can be increased due to frailty, elderly could be especially sensitive to the risk of hypoglycemia. Documentation of the total number of hypoglycemia is a relevant objective to really appreciate the potential impact of SUs in the Canadian context.

The investigators propose a multicenter observational prospective study in order to study the incidence of hypoglycaemia measured by CGMS among patients with type 2 diabetes mellitus (T2DM) newly prescribed a SU. The investigators propose to perform a baseline testing (pre-initiation of the SU), at initiation (first week after the first dose of the SU) and after a 3 months follow-up of treatment, including medical history measures, quality of life and diabetes treatment satisfaction.

In patients with T2DM not at goal (A1c >7.0 mmol/L), and newly prescribed a SU, the objectives and hypotheses of the study are to estimate the incidence rate of hypoglycaemia as measured by continuous glucose monitoring system (CGMS) over a total of 3 weeks period following the initiation of the SU.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes according to Canadian Diabetes Association definition
* Initiation of a SU at baseline
* A1c: 7.0% to 10.0%
* Willing and able to comply with study procedures

Exclusion Criteria:

* Current or previous usage (during the last 3 months) of insulin or repaglinide
* Use of medication known to interfere with glucose metabolism
* Insulin requiring patient: catabolic state and/or ketonuria
* Currently using CGMS or within the last 3 months
* Recent severe hypoglycemia (<3 months)
* Pregnancy or breast-feeding
* Limited life expectancy, high level of functional dependency, extensive coronary disease at high risk of short term ischemic events or multiple major co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM not at goal (A1c >7.0 mmol/L), and newly prescribed a SU
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Total incidence rate of hypoglycemia episode | One week after initiation of the SU
Total incidence rate of hypoglycemia episode | One week at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD,PhD, Principal Investigator — IRCM
Locations (2):
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Institut de recherches cliniques de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided